CLINICAL TRIAL: NCT06892093
Title: Efficacy and Safety of Probiotics Versus Standard Care in Preventing Diarrhea Induced by Neratinib in Breast Cancer Patients: A Prospective Randomized Controlled Clinical Trial
Brief Title: Probiotics for Prevention of Neratinib-Induced Diarrhea in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Jiangnan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSKY-2025-105-02
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-03

CONDITIONS: HER2-positive Breast Cancer; Diarrhea Caused by Drug; Neratinib
Keywords: Neratinib; Probiotics; Diarrhea; Breast Cancer
MeSH Terms: conditions — Diarrhea; Breast Neoplasms | interventions — Probiotics; Loperamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotics + Neratinib + Loperamide (Experimental)
  Interventions: Dietary Supplement: Probiotics; Drug: Loperamide
- Placebo + Neratinib + Loperamide (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo; Drug: Loperamide

INTERVENTIONS:
Dietary Supplement: Probiotics — Participants in this group will receive a daily dose of probiotics as an adjunct to standard Neratinib therapy. The probiotics will be administered orally as a granule formulation dissolved in water, for a total duration of 6 weeks (two treatment cycles). Loperamide will be administered prophylactically according to the FDA-recommended schedule to prevent Neratinib-associated diarrhea. The aim is to assess the efficacy of probiotics in reducing Neratinib-induced diarrhea and improving quality of life.
  Arms: Probiotics + Neratinib + Loperamide
Dietary Supplement: Placebo — Participants in this group will receive a daily dose of a placebo that is identical in appearance, taste, and administration method to the probiotic granules, in addition to standard Neratinib therapy. The placebo will be administered orally as a granule formulation dissolved in water, for a total duration of 6 weeks. Loperamide will also be administered prophylactically to all participants in accordance with FDA recommendations. This group will serve as a control to evaluate the true effect of probiotics on Neratinib-induced diarrhea.
  Arms: Placebo + Neratinib + Loperamide
Drug: Loperamide — All participants will receive prophylactic loperamide to reduce the risk of Neratinib-induced diarrhea. Loperamide will be administered according to the FDA-recommended schedule: 4 mg TID for the first 14 days of treatment, then 4 mg BID from Day 15 to Day 42. This intervention is implemented as a standard supportive therapy and not as a randomized variable.

SUMMARY:
This study aims to evaluate the efficacy and safety of probiotics for the prevention of diarrhea in patients with breast cancer receiving the tyrosine kinase inhibitor (TKI) Neratinib.

Study Design: This is a prospective, randomized controlled clinical trial. Participants will be randomly assigned to either a probiotics intervention group or a placebo-controlled group. Both groups will receive prophylactic loperamide according to the FDA-recommended dosing schedule for neratinib-associated diarrhea.

Primary Objective: To evaluate the efficacy of probiotics in reducing the incidence and severity of diarrhea in patients receiving Neratinib.

Secondary Objectives: This study will also investigate the effects of probiotics on gut microbiota composition and their potential impact on drug efficacy.

Study Duration: Enrollment is planned from August 2025 to June 2027 at Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University. Both the intervention and control groups will receive treatment for a total of six weeks (two cycles of three weeks each). No post-treatment observation period is included.

Eligibility Criteria: Participants must be diagnosed with HER2-positive breast cancer and scheduled to receive Neratinib. Exclusion criteria include patients with severe gastrointestinal disorders or recent probiotic consumption.

DETAILED DESCRIPTION:
Breast cancer patients treated with the tyrosine kinase inhibitor (TKI) Neratinib often experience severe diarrhea, leading to treatment interruptions, dose reductions, or discontinuation. Emerging evidence highlights the role of gut microbiota in drug metabolism and gastrointestinal toxicity. Probiotics have been proposed as a potential intervention to modulate gut microbiota and mitigate diarrhea; however, their efficacy in preventing Neratinib-induced diarrhea remains inconclusive.

This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the efficacy and safety of probiotics in preventing diarrhea in HER2-positive breast cancer patients receiving Neratinib. The study will also explore the impact of probiotics on gut microbiota composition and potential microbiome-mediated mechanisms that may enhance treatment adherence and therapeutic outcomes.

Participants will be randomly assigned in a 1:1 ratio to either a probiotics group or a placebo group. Both groups will receive prophylactic loperamide in accordance with the dosing schedule recommended by the U.S. Food and Drug Administration (FDA) for the prevention of Neratinib-associated diarrhea, ensuring consistency with the approved prescribing information.

Participants will receive treatment for a total of six weeks, corresponding to two treatment cycles.

Metagenomic sequencing and targeted metabolomics will be performed on stool samples to investigate gut microbial composition and metabolic changes. Additional analyses will assess the association between gut-derived metabolites and immune cell activation, aiming to elucidate potential interactions among gut microbiota, metabolites, and immune responses.

Sun Yat-sen Memorial Hospital will serve as the coordinating center for this planned multicenter trial. Currently, it is the only active site, and additional participating centers will be added progressively as they are initiated.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria:

1. Female patients aged ≥18 years, diagnosed with HER2-positive breast cancer.
2. Scheduled to receive Neratinib therapy (monotherapy or in combination), based on clinical guidelines.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, with an expected survival of at least 3 months.
4. Left ventricular ejection fraction (LVEF) ≥ 50%.
5. Resolution of any prior treatment-related toxicity to Grade ≤1 (per CTCAE v5.0), with AST and ALT ≤ 2.5 × the upper limit of normal (ULN), and total bilirubin ≤ 1.5 × ULN.
6. Adequate bone marrow function, defined as:

   White blood cell count ≥ 3.0 × 10⁹/L Neutrophil count ≥ 1.5 × 10⁹/L Platelet count ≥ 100 × 10⁹/L Hemoglobin ≥ 90 g/L Serum creatinine ≤ 1.5 × ULN
7. No persistent gastrointestinal symptoms, such as hematochezia, chronic constipation, or abdominal pain.
8. No evidence of structural gastrointestinal abnormalities confirmed by gastroscopy or other relevant examinations.

Exclusion Criteria

Participants will be excluded if they meet any of the following criteria:

1. Conditions that significantly impair swallowing, digestion, or gastrointestinal drug absorption.
2. History of chronic gastrointestinal diseases, including but not limited to inflammatory bowel disease (IBD), gastrointestinal tumors, or malabsorption syndromes.
3. Severe cardiovascular diseases that may interfere with study treatment, including but not limited to:

   Life-threatening arrhythmias Advanced atrioventricular block Unstable angina Clinically significant pericardial disease Myocardial fibrosis Uncontrolled hypertension
4. Known hypersensitivity to any component of Neratinib, probiotics, placebo, or loperamide.
5. Prior participation in any clinical trial involving investigational drugs within 4 weeks prior to enrollment, or chronic use of medications that may induce constipation within 6 months.
6. Pregnant or lactating women, or those unwilling to use effective contraception during the study period.
7. Any medical, psychiatric, or social condition that, in the investigator's judgment, could compromise the safety of the participant, interfere with study participation, or confound the study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade ≥3 Diarrhea | Up to 6 weeks
  The incidence of grade 3 or higher diarrhea during the 6-week treatment period, assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Incidence of Any Grade Diarrhea | Up to 6 weeks
  The incidence of diarrhea of any grade during the 6-week treatment period, assessed according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Duration of First Episode of Grade 3 Diarrhea | Up to 6 weeks
  The duration (in days) of the first episode of grade 3 diarrhea experienced by participants during the 6-week treatment period, assessed using the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Duration is defined from onset to recovery (downgrade to grade ≤2).
Proportion of Participants Hospitalized Due to Diarrhea | Up to 6 weeks
  The proportion of participants who require hospitalization due to diarrhea-related complications during the treatment period.
Loperamide Usage Patterns | Up to 6 weeks
  Frequency, total dosage, and compliance of loperamide use during the treatment period, including any dose modifications or discontinuation. Data will be collected through medication records and patient diaries.
Change from Baseline in Overall Quality of Life Assessed by EORTC QLQ-C30 | Baseline, Weeks 2, 4, and 6 (End of Study)
  Changes in quality of life assessed using the EORTC QLQ-C30 questionnaire. The tool evaluates overall health status and functioning, including physical, role, emotional, cognitive, and social domains. Higher scores in functional and global health scales indicate better quality of life, while higher scores in symptom scales indicate greater symptom burden.
Change from Baseline in Diarrhea-Related Quality of Life Assessed by FACT-D | Baseline, Weeks 2, 4, and 6 (End of Study)
  Changes in diarrhea-related quality of life assessed using the FACT-D subscale of the Functional Assessment of Cancer Therapy system. This tool specifically evaluates the severity and impact of diarrhea symptoms on patients' daily life and well-being. Higher scores indicate fewer symptoms and better diarrhea-related quality of life.
Incidence of Treatment-Related Adverse Events (AEs) | Up to 6 weeks
  The incidence of treatment-related adverse events (AEs) in participants receiving probiotics plus Neratinib versus the control group. AEs, including nausea, allergic reactions, and other related symptoms, will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Incidence of Serious Adverse Events (SAEs) | Up to 6 weeks
  The incidence of serious adverse events (SAEs) associated with probiotics or Neratinib treatment. SAEs, including severe allergic reactions, life-threatening complications, or hospitalizations, will be recorded and summarized to assess potential safety concerns.
Rate of Treatment Discontinuation Due to Adverse Events | Up to 6 weeks
  The proportion of participants who discontinue Neratinib treatment due to adverse events. The outcome will compare discontinuation rates between the probiotic and placebo groups to evaluate tolerability.

OTHER OUTCOMES:
Gut Microbiota Composition Changes | Baseline, Week 3, and Week 6
  Analysis of stool samples collected at baseline, week 3, and week 6 to assess changes in gut microbiota composition in response to probiotic intervention. The goal is to determine whether probiotics modulate the intestinal microbiota and exert a protective effect against Neratinib-associated diarrhea.
Correlation Analysis of Gut Microbiota-Metabolite-Immune Axis | Baseline, Week 3, and Week 6
  Integrated analysis of gut microbiota composition, blood and gut microbial metabolites, and immune response markers. This study aims to explore potential mechanistic links between gut microbiota, metabolite changes, and immune function.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Tumor Center, Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China